CLINICAL TRIAL: NCT01823627
Title: Pulmonary Disease in a Psychiatric Inpatient Population, a Screening Study
Brief Title: Pulmonary Disease in a Psychiatric Inpatient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psykiatrien Syd (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Principal Investigator, Nicolai Stig Renstrøm, 1.Reservelæge, Psykiatrien Syd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-322
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: COPD; Psychiatric inpatient; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spirometry with reversibility test (Other): Spirometry with reversibility test
  Interventions: Procedure: Spirometry with reversibility test

INTERVENTIONS:
Procedure: Spirometry with reversibility test — Spirometry with reversibility test and CATest questionaire. following will be measured FEV1 L/s FVC L/s FEV1/FVC ration
  Other Names: MicroLoop handheld transportable spirometer

SUMMARY:
Purpose: Patients with mental health disorders have a reduced life expectancy, compared to the general population. The shorter life expectancy is caused by natural and unnatural death. In general, patients with a mental disorder tend to have a more unhealthy lifestyle, than the general population, characterized by e.g. lack of exercise and smoking.

Hypothesis

Chronic obstructive pulmonary disease (COPD) is underdiagnosed in psychiatric inpatients There is a higher prevalence of COPD in psychiatric inpatients compared to the general population Screening of patients with one respiratory symptom and a smoking history, has the same sensitivity regarding to diagnosis of COPD, as screening all patients with a smoking history

Method:

80 psychiatric inpatients will undergo spirometry with reversibility test and COPD Assessment Test (CATest). Furthermore, patient history regarding respiratory symptoms and smoking will be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in Psykiatrien Syd, Region Zealand, ward S1,S2,S3,S4,S5,S6
* Admission time over 48 hours

Exclusion Criteria:

* Patients who is not able to perform spirometry due to their psychiatric condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Tiffeneau index | at enrollment
  - FEV1/FVC ratio

SECONDARY OUTCOMES:
forced vital capacity | at enrollment
  FVC L/s
Forced expiratory volume in 1 second | at enrollment
  FEV1 L

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Renstrom, Principal Investigator — Psykiatrien Syd
Locations (1):
- Psyciatrien Syd, Region Zealand, Vordingborg, Denmark

IPD SHARING:
Plan to Share IPD: No